CLINICAL TRIAL: NCT05823506
Title: Efficacy and Safety of Focused Shockwave Therapy Plus Tadalafil vs Tadalafil Alone in Patient With Erectile Dysfunction: Randomized Controlled Trial
Brief Title: Efficacy and Safety of Focused Shockwave Therapy Plus Tadalafil vs Tadalafil Alone in Patient With Erectile Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Saint Petersburg State University, Russia (Other)
Responsible Party: Principal Investigator, Gleb Kovalev, The head of outpatient urology department, phD, Saint Petersburg State University, Russia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESWT_tadalafil_in_ED
Record Dates: First submitted 2023-04-10; First posted 2023-04-21 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Phosphodiesterase 5 Inhibitors; Tadalafil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medication group (Active Comparator): PDE5 inhibitor tadalafil in dosage 5 mg daily by 1 month
  Interventions: Drug: PDE5 inhibitor (tadalafil)
- Combination group (Experimental): PDE5 inhibitor tadalafil in dosage 5 mg daily by 1 month plus Device BTL-6000 fSWT: 6 sessions with EFD 0,09 mJ/mm2 by 5000 impulses per session in 5 points in corpora cavernosa penis
  Interventions: Combination Product: PDE5 inhibitor (tadalafil) and BTL-6000 fSWT; Drug: PDE5 inhibitor (tadalafil)

INTERVENTIONS:
Combination Product: PDE5 inhibitor (tadalafil) and BTL-6000 fSWT — The mechanism of low-intensity shockwave therapy in patients with ED based on the effect on the endothelium of the cavernous arteries, the release of NO and the enhancement of vascularization due to release of angiogenic factors.
  Arms: Combination group
Drug: PDE5 inhibitor (tadalafil) — Tadalafil improves erectile function by inhibiting PDE5 isoenzyme, thereby blocking cGMP degradation. As a result, the PDE5 inhibitors act synergistically with NO to markedly increase the levels of cGMP, which in the presence of sexual stimulation, lead to an erection. In the absence of sexual stimulation, NO is not released locally and the PDE5 inhibitors do not affect the penis. Thus, sexual stimulation is needed to initiate the erectile mechanism for the PDE5 inhibitors to take effect.

SUMMARY:
The goal of this trial is that using tadalafil plus low-intensity extracorporeal shockwave therapy (li-ESWT) is more effective than using tadalafil alone in improving erection rigidity and sexual function. The efficacy of the combination of li-ESWT and tadalafil has been confirmed by a number of studies, including in patients after radical prostatectomy. However, this method is still not a "first-line" method in young primary patients and its benefits in combination with drugs for these patients are not obvious.

The investigators assume that the combination of tadalafil plus low-intensity extracorporeal shockwave therapy (li-ESWT) will improve the subjective state of patients assessed by points of validated questionnaires and Number of successful intercourse per week.

DETAILED DESCRIPTION:
The aim of the study is to test the hypothesis that using tadalafil plus shockwave in primary patient with ED treatment in more effective in improving erection rigidity and sexual function, then using tadalafil alone.

ELIGIBILITY:
Inclusion Criteria:• Age 20 to 45;

* Married or have had a permanent sex partner for at least 3 months;
* IIEF-5 questionnaire scores below 20

Exclusion Criteria:

* History of previous use of PDE-5 inhibitors or fSWT;
* Patients with diabetes mellitus;
* Patients after the radical prostatectomy or major pelvic surgery;
* Patients with a confirmed neurological disease that may have caused the ED (Multiple Sclerosis, Parkinson's Disease, spinal cord injury);
* Patients with contraindications to the use of PDE-5 inhibitors and/or fSWT;

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — because the study examines the effects of PDE-5 inhibitors or fSWT on erectile function in men
Enrollment: 36 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
IIEF-5 | 60 days
  IIEF-5 (International Index of Erectile Function-5) is validated erectile function assessment questionnaire. The possible scores for the IIEF-5 range from 5 to 25, with lower values representing poorer sexual function.

SECONDARY OUTCOMES:
PGI-I | 14 days,30 days, 60days.
  The Patient Global Imression of Improvement (PGI-I) is a global index that may be used to rate the response of a condition to a therapy. This is a transition scale that is a single question asking the patient to rate their urinary tract condition now, as compared with how it was prior to before beginning treatment on a scale from 1-Very much better to 7-Very much worse.
Likert scale (7-point preferably) satisfaction questionnaire | 14 days,30 days, 60days.
  Likert Scale questions offer a range of answer options from either end of the spectrum for the respondents to choose from, where 1-extremely dissatisfied, 7- extremely satisfied
Therapy comfort survey | 14 days,30 days, 60days.
  Modified scale indicating how comfort patients feel about therapy, where 1is totally uncomfortable, and 7 is very comfortable.
Number of successful intercourse per week | 14 days,30 days, 60days.
  Number of successful intercourse per week

CONTACTS AND LOCATIONS:
Locations (1):
- SBPSU, Saint Petersburg, Russia